CLINICAL TRIAL: NCT06128603
Title: Analysis of Intraoperative Bleeding Characteristics in Laparoscopic Pancreaticoduodenectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinrui Zhu，MD (Other)
Responsible Party: Sponsor-Investigator, Xinrui Zhu，MD, attending doctor, West China Hospital
Organization: West China Hospital (Other)
Other Study IDs: 2023-1663-1
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Laparoscopic Pancreaticoduodenectomy
Keywords: laparoscopic pancreaticoduodenectomy; intraoperative bleeding; OSATS scores; short-time outcomes
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LPD group: Cases who had underwent laparoscopic pancreaticoduodenectomy
  Interventions: Procedure: laparoscopic pancreaticoduodenectomy

INTERVENTIONS:
Procedure: laparoscopic pancreaticoduodenectomy — laparoscopic pancreaticoduodenectomy was performed for periampullary benign and malignant diseases. Besides, the surgical video was recorded.

SUMMARY:
In this study, we analyze the common bleeding characteristics in laparoscopic pancreaticoduodenectomy by reviewing and annotating bleeding information from previous surgical videos as well as surgical operation OSATS technique scores. From there, we reflect on the correlation between surgical operating technique and intraoperative bleeding, as well as on the correlation between intraoperative bleeding and short-term postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* the surgical video is complete including the resection and reconstruction phases

Exclusion Criteria:

* the surgical video is not complete
* the cases combined with resection and reconstruction of mesentericoportal vein

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients underwent laparoscopic pancreaticoduodenectomy for periampullary benign and malignant diseases.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-25 (Estimated)

PRIMARY OUTCOMES:
intraoperative bleeding characteristics | intraoperatively
  Bleeding characteristics include cause of bleeding, site of bleeding, size of bleeding, method of hemostasis, duration of hemostasis, and outcome of hemostasis. These would be obtained by reviewing and labeling laparoscopic pancreaticoduodenectomy surgical videos.

SECONDARY OUTCOMES:
OSATS scores | intraoperatively
  Scoring laparoscopic pancreaticoduodenectomy operations using the OSATS Surgical Operative Technique Rating Scale
textbook outcome | 3 months postoperatively
  The textbook outcome was defined as the absence of all six individual outcomes: clinically relevant postoperative pancreatic fistula, post-pancreatectomy hemorrhage, bile leak, severe complications (Clavien-Dindo≥3), readmission, and mortality within 30 days postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No